CLINICAL TRIAL: NCT05636371
Title: Impact of WRitten Communication on the ICU Team Experience
Brief Title: Written Communication in the Intensive Care Unit
Acronym: WRITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22092704-IRB01
Record Dates: First submitted 2022-10-31; First posted 2022-12-05 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Communication; Satisfaction, Patient; Burnout
MeSH Terms: conditions — Communication; Patient Satisfaction; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Written Communication (Experimental): ICU care providers will initiate the process for providing written communication to families. Study investigators will facilitate the creation and distribution of written communication
  Interventions: Other: Written Communication

INTERVENTIONS:
Other: Written Communication — Written patient care updates provided to families of ICU patients each day

SUMMARY:
The goal of this study is to compare the experience of intensive care unit (ICU) families and care providers before and after the implementation of an approach whereby clinicians initiate written communication with families

The main questions it aims to answer are

1. Is ICU care-provider initiated written communication feasible and acceptable to participants?
2. Does ICU care-provider initiated written communication affect the experience of families and care providers?

Participants will complete surveys and participate in interviews during a 3 month pre-implementation phase and a 3 month post-implementation phase

ELIGIBILITY:
Inclusion criteria (family members or surrogates)

• Self-identify as one of the patient's decision makers

Exclusion criteria (family members or surrogates)

* Cannot read or understand English
* Unwilling to participate in study procedures

Inclusion criteria for care providers (physicians, physician assistants, and nurses)

• Work during the day shift

Exclusion criteria for care providers (physicians, physician assistants, and nurses)

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Family Inpatient Communication Survey (FICS) | 5 days after ICU admission
  The Family Inpatient Communication Survey (FICS) is a 30-item survey measuring of the quality of communication with the treatment team from the perspective of families of hospitalized patients. Items on this survey measure the informational and emotional aspects of communication, and each item of this survey is rated on a 5-point Likert scale from strongly agree to strongly disagree. The FICS has been validated in a study of 350 surrogates of hospitalized adults demonstrating the high internal reliability, predictive validity, and high item completion rates of this survey.
Family Inpatient Communication Survey (FICS) | 10 days after ICU admission
  The Family Inpatient Communication Survey (FICS) is a 30-item survey measuring of the quality of communication with the treatment team from the perspective of families of hospitalized patients. Items on this survey measure the informational and emotional aspects of communication, and each item of this survey is rated on a 5-point Likert scale from strongly agree to strongly disagree. The FICS has been validated in a study of 350 surrogates of hospitalized adults demonstrating the high internal reliability, predictive validity, and high item completion rates of this survey.
Nurse-Physician Collaboration Scale (NPCS) | 3 months before the intervention
  The Nurse-Physician Collaboration Scale (NPCS) is a 27-item survey measuring the level of collaboration between nurses and physicians based on three categories: joint participation in the decision-making process, the sharing of patient information, and cooperativeness.Items on this survey are rated on a 5-point scale with responses ranging from always to never. The NPCS has been validated in a study of 446 physicians and 1217 nurses at 27 hospitals.
Nurse-Physician Collaboration Scale (NPCS) | 3 months after the intervention
  The Nurse-Physician Collaboration Scale (NPCS) is a 27-item survey measuring the level of collaboration between nurses and physicians based on three categories: joint participation in the decision-making process, the sharing of patient information, and cooperativeness.Items on this survey are rated on a 5-point scale with responses ranging from always to never. The NPCS has been validated in a study of 446 physicians and 1217 nurses at 27 hospitals.
Maslach Burnout Inventory (MBI) | 3 months before the intervention
  The Maslach Burnout Inventory (MBI) is a 22-item survey measuring symptoms of burnout. The MBI has been validated for a variety of professions. The MBI has been used in past studies in the ICU to evaluate the level of burnout present among critical care clinicians and to assess for the effectiveness of interventions attempting to alleviate the degree of burnout syndrome. This survey examines the participant's perception of their work, physical and emotional exhaustion, sense of personal accomplishment, and degree of depersonalization. Items are presented as single statements, such as "I feel worn out at the end of a working day," and are rated on a scale of 0 to 6 with 0 being "never" and 6 being "every day."
Maslach Burnout Inventory (MBI) | 3 months after the intervention
  The Maslach Burnout Inventory (MBI) is a 22-item survey measuring symptoms of burnout. The MBI has been validated for a variety of professions. The MBI has been used in past studies in the ICU to evaluate the level of burnout present among critical care clinicians and to assess for the effectiveness of interventions attempting to alleviate the degree of burnout syndrome. This survey examines the participant's perception of their work, physical and emotional exhaustion, sense of personal accomplishment, and degree of depersonalization. Items are presented as single statements, such as "I feel worn out at the end of a working day," and are rated on a scale of 0 to 6 with 0 being "never" and 6 being "every day."

SECONDARY OUTCOMES:
The Acceptability, Appropriateness and Feasibility of Intervention Survey (AIM, IAM and FIM) | 3 months after the intervention
  Care providers will complete this 12-item psychometric assessment. Implementation science researchers have established the benchmarks and acceptance of this scale.
The Post Study System Usability Questionnaire (PSSUQ) | 3 months after the intervention
  The Post Study System Usability Questionnaire (PSSUQ) is a 16-item PSSUQ survey that measures the acceptance of new technology. PSSUQ measures perception of information quality, interface quality, and overall intervention usefulness. Lewis et al have published on the high internal validity and sensitivity of this scale since 1992.
The User Experience Questionnaire (UEQ) | 3 months after the intervention
  The User Experience Questionnaire (UEQ) is a 8-item scale to measure the overall user experience of the family member(s) who used the communication intervention. The UEQ measures user experience on items including attractiveness, perspicuity, efficiency, dependability, stimulation, and novelty. UEQ has high internal validity and has been benchmarked across numerous usability and user experience evaluation studies.

OTHER OUTCOMES:
Qualitative analysis | 3 months after the intervention
  Semi-structured interviews with participants will be coded and examined using thematic content analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Greenberg JA, Basapur S, Quinn TV, Bulger JL, Schwartz NH, Oh SK, Ritz EM, Glover CM, Shah RC. Daily Written Care Summaries for Families of Critically Ill Patients: A Randomized Controlled Trial. Crit Care Med. 2022 Sep 1;50(9):1296-1305. doi: 10.1097/CCM.0000000000005583. Epub 2022 May 23. PMID 35607975
- [Background] Grant M. Resolving communication challenges in the intensive care unit. AACN Adv Crit Care. 2015 Apr-Jun;26(2):123-30. doi: 10.1097/NCI.0000000000000076. PMID 25898880
- [Background] Kerlin MP, McPeake J, Mikkelsen ME. Burnout and Joy in the Profession of Critical Care Medicine. Crit Care. 2020 Mar 24;24(1):98. doi: 10.1186/s13054-020-2784-z. PMID 32204724
- [Background] Wright AA, Katz IT. Beyond Burnout - Redesigning Care to Restore Meaning and Sanity for Physicians. N Engl J Med. 2018 Jan 25;378(4):309-311. doi: 10.1056/NEJMp1716845. No abstract available. PMID 29365301